CLINICAL TRIAL: NCT05838833
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Clinical Trial to Evaluate the Efficacy and Safety of INV-001 Administration for the Prevention of Scar After Thyroidectomy
Brief Title: Ointment to Prevent Scar After Thyroidectomy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Innovo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: INV001-01
Record Dates: First submitted 2023-03-29; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Scar
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose (Experimental): low dose ointment
  Interventions: Drug: INV-001
- High dose (Experimental): high dose ointment
  Interventions: Drug: INV-001
- Placebo (Placebo Comparator): same ingredient with active drug except API
  Interventions: Drug: INV-001

INTERVENTIONS:
Drug: INV-001 — Patient will be assigned to one of three arms.

SUMMARY:
The goal of this study is to evaluate the efficacy and Safety of INV-001 administration for the prevention of scar after thyroidectomy.

Participants will be asked to apply ointment on their scar for 12 weeks.

DETAILED DESCRIPTION:
to evaluate the efficacy

-investigator check POSAS and VSS

ELIGIBILITY:
Inclusion Criteria:

* Patient who got thyroidectomy due to Thyroid cancer
* has scar longer than 3 cm

Exclusion Criteria:

* have history about Keloid or Hypertrophic scar
* have infection on surgical site

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Observer overall opinion of POSAS | 12 weeks
  POSAS POSAS: Patient Observer Scar Assessment Scale

SECONDARY OUTCOMES:
Observer overall opinion of POSAS | 3, 6 weeks
  POSAS: Patient Observer Scar Assessment Scale

CONTACTS AND LOCATIONS:
Overall Officials: Minjeong Kim, Master, Study Director — New Drug development Center
Locations (1):
- Innovo Therapeutics, Inc., Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided